CLINICAL TRIAL: NCT06285552
Title: Evaluation of the Comprehensive Family Support Program (PAIF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Gobierno de Cantabria (Unknown); Loyola University (Other); University of Jaen (Unknown)
Responsible Party: Principal Investigator, Victoria Hidalgo García, Principal Investigator, University of Seville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4792/0842
Record Dates: First submitted 2024-02-07; First posted 2024-02-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Parenting
Keywords: Positive parenting; Parenting competences; Program evaluation; Family functioning; Parenting practices; Effectiveness

STUDY DESIGN:
Intervention Model Description: The participants will be assigned to the manualized program according to the inclusion criteria. The comparison group will be composed of families in areas where the intervention is not available but with similar sociodemographic characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Parenting newborn (Experimental): Program aimed at community families with children enrolled in Early Childhood Care Centers (from 0 to 2 years old).
  Interventions: Behavioral: Positive parenting PAIF program
- Parenting Toddlers (Experimental): Program aimed at community families with children from 2 to 5 years old.
  Interventions: Behavioral: Positive parenting PAIF program
- Parenting Children (Experimental): Program aimed at community families with children from 6 to 12 years old.
  Interventions: Behavioral: Positive parenting PAIF program
- Parenting Adolescents (Experimental): Program aimed at community families with children from 12 to 18 years old.
  Interventions: Behavioral: Positive parenting PAIF program
- Active and Health Families (Experimental): Program aimed at targeted families due identified needs for healthy lifestyle habits
  Interventions: Behavioral: Positive parenting PAIF program
- Functional diversity Parenting (Experimental): Program aimed at targeted families whose children and/or adolescents exhibit functional diversity characteristics
  Interventions: Behavioral: Positive parenting PAIF program
- Control (No Intervention): Families that are not participating in any program as they live in a comparable area where any of the intervention is offered
- Parenting as as Father (Experimental): Program aimed at fathers from the community population
  Interventions: Behavioral: Positive parenting PAIF program

INTERVENTIONS:
Behavioral: Positive parenting PAIF program — Psychoeducational intervention in a group format driven by a practitioner with 6 to 12 sessions where caregivers learn parenting competences
  Arms: Active and Health Families; Functional diversity Parenting; Parenting Adolescents; Parenting Children; Parenting Toddlers; Parenting as as Father; Parenting newborn

SUMMARY:
The goal of this study is to evaluate the effectiveness of positive parenting programs targeted to parents of toddlers, children and adolescents carried out in Cantabria (Spain).

We will collect information from the participants before the intervention, in the last session of the program and some months after, to verify if there have been some changes in the family dynamics of these parents, and if these changes continue after some time. Besides, we will compare these results with information from other families that are not taking part in the program. The main caregivers of the participating families and the practitioners in charge of the intervention will provide the information for the study.

We expect that families participating in the programs will improve their parenting competencies and their family dynamics, and that these change will stay after the program.

DETAILED DESCRIPTION:
A quasi-experimental design will be followed, with three evaluation moments (pretest, posttest and follow-up) and with a non-randomized comparison group.

The positive parenting programs will be advertised by social media, schools and high schools. The participants will be parental figures interested in joining these programs.

The participants will answer a series of questionnaires by an app, where they will give information related to sociodemographic data and parenting competencies. The app will not allow the participants to leave any question with no answer or with an incorrect answer.

To analyze the data, we will use the softwares Mplus and Statistical Package for the Social Sciences (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* Being caregiver of at least one child under 18 years of age
* The child to be in the developmental stage appropriate for the corresponding arm
* If participating in a targeted program, meet the requirements: (1) be a father; (2) presenting bad health habits in the family according the evaluation of the pediatrician
* Motivated to improve parenting competences

Exclusion Criteria:

* Not having sufficient command of the Spanish language to be able to communicate
* Experience family crisis that prevent for participating in a group intervention
* Experience mental health issue that prevent for participating in a group intervention

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Perception of the parental role | Pretest, immediately posttest and 6 month follow-up
  Me as a Parent Scale (MaaP), rated on a 5-point Likert-type scale ranging from 1 to 5. Higher scores mean a better outcome.
Parenting practices (Authoritative parenting style: Warmth and Support, Reasoning/Induction, Democratic Participation) | Pretest, immediately posttest and 6 month follow-up
  Parenting Styles and Dimensions Questionnaire - Short version (PSDQ-Short version), rated on a 5-point Likert-type scale ranging from 1 to 5. Higher scores mean a better outcome.
Parenting practices (Overreactivity and Laxness) | Pretest, immediately posttest and 6 month follow-up
  Parenting Scale - Short version (PS), rated on a 7-point Likert-type scale ranging from 1 to 7. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Satisfaction with the intervention | Immediately Posttest
  Client Satisfaction Questionnaire (CSQ-4), rated on a 4-point Likert-type scale ranging from 1 to 4. Higher scores mean a better outcome.
Children adjustment | Pretest, immediately posttest and 6 month follow-up
  Kidscreen-10, rated on a 5-point Likert-type scale ranging from 1 to 5. Higher scores mean a better outcome.
Social support | Pretest, immediately posttest and 6 month follow-up
  Ad hoc questionnaire, with 3 items rated on a 5-point Likert-type scale ranging from 1 = Nothing to 4 = A lot ("I feel supported as a father/mother). Higher scores mean a better outcome.
Satisfaction with Family Life | Pretest, posttest and follow-up
  Satisfaction with Family Life Scale (SWFLS), rated on a 7-point Likert-type scale ranging from 1 to 7. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Consejería de Inclusión Social, Juventud, Familias E Igualdad, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No
The project is framed in an agreement with the Govern of Cantabria and the researchers have no authorization for sharing individual participant data.

REFERENCES:
- [Background] Hamilton, V., Matthews, J. & Crawford, S. (2015). Development and preliminary validation of a parenting self-regulation scale: "Me as a Parent". Journal of Child & Family Studies. 24(10), 2853-2864. https://doi.org/10.1007/s10826-014-0089-z
- [Background] Robinson, C. C., Mandleco, B., Olsen, S. F., & Hart, C. H. (1995). Authoritative, Authoritarian, and Permissive Parenting Practices: Development of a New Measure. Psychological Reports, 77(3), 819-830. https://doi.org/10.2466/pr0.1995.77.3.819
- [Background] Reitman D, Currier RO, Hupp SD, Rhode PC, Murphy MA, O'Callaghan PM. Psychometric characteristics of the Parenting Scale in a head start population. J Clin Child Psychol. 2001 Dec;30(4):514-24. doi: 10.1207/S15374424JCCP3004_08. PMID 11708239
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Ramon B. Zabriskie & Peter J. Ward (2013) Satisfaction With Family Life Scale, Marriage & Family Review, 49:5, 446-463, DOI: 10.1080/01494929.2013.768321
- See also: Website of the instrument Kidscreen-10 — https://www.kidscreen.org/english/questionnaires/kidscreen-10-index/